CLINICAL TRIAL: NCT07123129
Title: An Open-label, Multicenter Phase I Clinical Study of SHR-7782 Injection in the Treatment of Advanced Malignant Cancer
Brief Title: A Trial of SHR-7782 for Treatment of Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-7782-101
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-7782 Group (Experimental)
  Interventions: Drug: SHR-7782 Injection

INTERVENTIONS:
Drug: SHR-7782 Injection — SHR-7782 injection.

SUMMARY:
The main objective of this study is to evaluate the effectiveness and safety of SHR-7782 for participants with advanced malignant cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Participate in the study voluntarily, sign the informed consent form.
2. Subjects were able to provide primary or metastatic cancer samples.
3. At least one measurable lesion (RECIST version 1.1).
4. ECOG 0~1.
5. With adequate organ functions.
6. Expected survival time ≥ 12 weeks.

Exclusion Criteria:

1. With untreated brain metastasis or active central nervous system tumor metastases.
2. Imaging shows that the tumor invades large blood vessels or has unclear boundaries with blood vessels.
3. Patients with other malignant tumors in the past or at the same time.
4. Patients with clinical symptoms, uncontrolled, or moderate or above pleural effusion, pericardial effusion, or peritoneal effusion.
5. Patients with a history of interstitial pneumonia or interstitial lung disease or non-infectious pneumonia requiring steroid treatment.
6. With poorly controlled or severe cardiovascular disease.
7. Bleeding events of NCI-CTCAE v5.0 grade ≥ 2 occurred within 1 month before the first medication.
8. Subjects who had a serious infection within 1 month before the first medication.
9. History of immunodeficiency.
10. Known allergy to any component of the SHR-7782 product.
11. According to the researcher's judgment, there are other factors that may affect the research results or cause the research to be terminated midway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | Up to 21 days.
Maximum Tolerated Dose (MTD) | Up to 6 months.
Recommended Phase II Dose (RP2D) | Up to 21 days.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) assessed by the investigator according to RECIST 1.1 criteria | Up to approximately 24 months.
Duration of Response (DoR) assessed by the investigator according to RECIST 1.1 criteria | Up to approximately 24 months.
Disease Control Rate (DCR) assessed by the investigator according to RECIST 1.1 criteria | Up to approximately 24 months.
Progression Free Survival (PFS) assessed by the investigator according to RECIST 1.1 criteria | Up to approximately 24 months.
Overall Survival (OS) | Up to approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided